CLINICAL TRIAL: NCT06932562
Title: A Randomized, Open-Label, Controlled Phase 3 Study of Comparing Daratumumab, Lenalidomide and Dexamethasone Induction Followed by Linvoseltamab Versus Continued Daratumumab, Lenalidomide, and Dexamethasone in Newly Diagnosed Transplant Ineligible Multiple Myeloma Patients
Brief Title: A Study to Learn How Safe and How Well Linvoseltamab Works Compared to Standard Treatment in Adult Patients With Multiple Myeloma Who Are Not Eligible for Transplant
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: European Myeloma Network B.V. (Network)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMN39; 2024-519827-16-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma (MM); Transplant ineligible; Newly diagnosed; Linvoseltamab; BCMA X CD3 bispecific antibody; CD38 antibody; Lenalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control arm DRd (Active Comparator)
  Interventions: Drug: Daratumumab; Drug: Lenalidomide; Drug: Dexamethasone
- Experimental Arm DRd+ linvolsetamab (Experimental)
  Interventions: Drug: Linvoseltamab; Drug: Daratumumab; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Linvoseltamab — Administered per the protocol
  Other Names: REGN5458
  Arms: Experimental Arm DRd+ linvolsetamab
Drug: Daratumumab — Administered per the protocol
Drug: Lenalidomide — Administered per the protocol
Drug: Dexamethasone — Administered per the protocol

SUMMARY:
This study is researching an experimental drug called linvoseltamab. The study is focused on participants with newly diagnosed multiple myeloma (NDMM) who are ineligible for autologous stem cell transplantation (transplant-ineligible).

The main purpose of this study is to compare the effect and safety of linvoseltamab with the effect and safety of the standard treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have confirmed diagnosis of symptomatic MM per IMWG criteria.
2. Participants must not be considered a candidate for high-dose chemotherapy (HDT) and ASCT, as described in the protocol.
3. Participants must have measurable disease as defined in the protocol.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
5. Participants must have clinical laboratory values within a prespecified range.

Exclusion Criteria:

1. International Myeloma Working Group Frailty Index of 2 with the exception of participants who have a score of 2 based on age alone.
2. Participants who defer transplant due to personal preference.
3. Participants with non-secretory MM, active plasma cell leukemia, known light-chain (AL) amyloidosis in the presence of a concurrent diagnosis of myeloma, any other form of amyloidosis, Waldenström macroglobulinemia, or known POEMS syndrome.
4. Any prior therapy for monoclonal gammopathy of undetermined significance (MGUS), smoldering multiple myeloma (SMM), or MM, with the exception of:

   * focal radiation and/or
   * a short course of corticosteroids as defined in the protocol.
5. Participants who have received or are receiving any investigational agent or cell therapy with known or suspected activity against MM
6. Participants who have known central nervous system (CNS) or meningeal involvement with MM or known or suspected progressive multifocal leukoencephalopathy (PML), a history of a neurocognitive condition or CNS movement disorder, OR a history of seizure, transient ischemic attack (TIA), stroke or seizure within 12 months prior to study C1D1.
7. Participants who have uncontrolled intercurrent illness.
8. Known contraindications to the use of daratumumab or lenalidomide per local prescribing information.
9. History of allogeneic hematopoietic stem cell transplantation or solid organ transplant at any time.

NOTE Other protocol defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-12-23 (Actual); Primary Completion 2036-12 (Estimated); Study Completion 2036-12 (Estimated)

PRIMARY OUTCOMES:
Minimal Residual Disease (MRD) | up to 11 years
  Minimal Residual Disease (MRD) negative Complete Remission (CR) status at 10^-5 per International Myeloma Working Group (IMWG) criteria
MRD negative CR status by BICR | up to 11 years
  MRD negative CR status at 10^-5 as determined by the Blinded Independent Central Review (BICR)
Progression Free Survival (PFS) per IMWG criteria | up to 11 years
  defined as the time from the date of randomization until the first occurrence of disease progression or death from any cause, whichever occurs earlier, where disease progression is determined per IMWG criteria.
PFS as determined by BICR | up to 11 years
  defined as the time from the date of randomization until the first occurrence of disease progression or death from any cause, whichever occurs earlier, where disease progression is determined per by BICR.

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 11 years
  Overall Survival (OS), measured from the date of from randomization to the date the subject's death
Objective Response (OR) of Complete Response (CR) | up to 11 years
  To compare the proportion of patients who achieve an objective response per International Myeloma Working Group (IMWG) response criteria between the two study arms for Complete Response (CR) or better
OR of Very Good Partial Response (VGPR) | up to 11 years
  To compare the proportion of patients who achieve an objective response per International Myeloma Working Group (IMWG) response criteria between the two study arms for VGPR or better
OR of Partial Response (PR) | up to 11 years
  To compare the proportion of patients who achieve an objective response per International Myeloma Working Group (IMWG) response criteria between the two study arms for PR or better
Sustained MRD | up to 11 years
  Sustained MRD negative CR (sMRD) at 10^-5 per IMWG criteria
Duration of response (DOR) of stringent (s)CR | up to 11 years
  duration of response to best overall response of stringent sCR, per IMWG response criteria
Duration of response (DOR) of CR | up to 11 years
  duration of response to best overall response of CR, per IMWG response criteria
Duration of response (DOR) of VGPR | up to 11 years
  duration of response to best overall response of VGPR, per IMWG response criteria
Duration of response (DOR) of PR | up to 11 years
  duration of response to best overall response of PR, per IMWG response criteria
Time to response ≥CR | up to 11 years
  Time from randomization to objective response (≥CR) as per IMWG response criteria
Time to response ≥VGPR | up to 11 years
  Time from randomization to objective response (≥VGPR) as per IMWG response criteria
Time to response ≥PR | up to 11 years
  Time from randomization to objective response (≥PR) as per IMWG response criteria
Disease progression | up to 11 years
  Time to disease progression per IMWG response criteria
Incidence of TEAEs | up to 11 years
  Incidence of treatment emergent adverse events (TEAEs)
Severity of TEAEs | up to 11 years
  Severity of treatment emergent adverse events (TEAEs)
Serious Adverse Events | up to 11 years
  Incidence of Serious Adverse Events (SAE)
Concentrations of linvoseltamab | up to 11 years
  Concentrations of linvoseltamab in serum over time
Incidence antidrug antibodies | up to 11 years
  Incidence of antidrug antibodies (ADAs) to linvoseltamab
Titer of ADA | up to 11 years
  Titer of ADA to linvoseltamab
EORTC QLQ-C30 Global Health Status / Quality of Life | up to 11 years
  Change in European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30) The EORTC QLQ-C30 is a 30-item validated questionnaire developed to measure patient-reported quality of life using one global health status/quality of life (GHS/QoL) scale, 5 functioning scales (physical, role, emotional, cognitive, and social) ranging from from 1 = "very poor" to 7 = "excellent" and 9 symptom scales/items (fatigue, nausea/vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties) among patients with cancer, ranging from 1 = "not at all" to 4 = "very much" higher scores indicate higher symptom burden.
EORTC QLQ-C30 Physical Functioning (PF) | up to 11 years
  Change in European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire functioning scale Physical Functioning (PF). PF scale consist of 5 items, ranging from from 1 = "not at all" to 4 = "very much" higher scores indicate higher ("better") level of functioning
EORTC QLQ-C30 Role Functioning (RF) | up to 11 years
  Change in European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire functioning scale Role Functioning (RF). RF scale consist of 2 items, ranging from from 1 = "not at all" to 4 = "very much" higher scores indicate higher ("better") level of functioning
EORTC QLQ-C30 Pain | up to 11 years
  Change in European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire symptom scale Pain. Pain scale consist of 2 items, ranging from from 1 = "not at all" to 4 = "very much" higher scores indicate higher symptom burden
EORTC QLQ-C30 Fatigue | up to 11 years
  Change in European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire symptom scale Fatigue. Fatigue scale consist of 3 items, ranging from from 1 = "not at all" to 4 = "very much" higher scores indicate higher symptom burden
EQ-5D-5L VAS | up to 11 years
  Change in EuroQoL-5 Dimensions, 5-level Questionnaire (EQ-5D-5L) Visual Analogue Score (VAS) (EQ-5D-5L VAS).
  The EQ-5D-5L is a generic questionnaire that measures Health-Related Quality of Life (HRQoL) across 5 dimensions of health (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) across 5 levels (1= no problems, 2= slight problems, 3= some problems, 4= severe problems and 5= extreme problems), higher scores indicate lower health states And a visual analogue scale (VAS). VAS scale ranging from 0 = "worst" to 100 = "best" higher score indicate higher health status

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Mina, Principal Investigator — A.O.U. Città della Salute e della Scienza di Torino; Claudia Stege, Principal Investigator — Erasmus Medical Center
Locations (33):
- Australia (3):
  - Austin Hospital, Heidelberg
  - Nepean Cancer Centre, Kingswood
  - Sunshine Coast Health, Sunshine Coast
- Ordensklinikum Linz, Linz, Austria
- Czechia (4):
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - University Hospital Olomouc, Olomouc
  - Fakultni Nemocnice Ostrava, Ostrava
  - Fakultni Nemocnice Plzen, Pilsen
- Aarhus Universitetshospital, Aarhus, Denmark
- Estonia (2):
  - North Estonia Medical Centre Foundation, Tallinn
  - Tartu University Hospital, Tartu
- Kuopio University Hospital, Kuopio, Finland
- University Hospital of Würzburg, Würzburg, Germany
- Italy (7):
  - AOU Ospedali Riuniti di Ancona, Ancona
  - A.O.U. Careggi, Florence
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Meldola-Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.), Meldola
  - Azienda USL IRCCS Di Reggio Emilia, Reggio
  - Ospedale "Infermi" di Rimini, Rimini
  - I.R.C.C.S. Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
- Erasmus MC, Rotterdam, Netherlands
- Norway (3):
  - Stavanger University Hospital, Stavanger
  - St. Olavs hospital HF, Trondheim
  - Vestfold Hospital Trust, Tønsberg
- Portugal (2):
  - CHUC, Coimbra
  - Hospital da Luz Lisboa, Lisbon
- Spain (4):
  - Hospital Clinic De Barcelona - Myeloma and Amyloidosis Unit, Barcelona
  - Hospital Quirón Salud Madrid, Madrid
  - Hospital Universitario Marques De Valdecilla -Hematology and Hemotherapy Service, Santander
  - Hospital Universitario la Fe, Valencia, Valencia
- Switzerland (2):
  - Universitaetsspital Basel - Zentrum fur Hamato-Onkologie, Basel
  - Kantonsspital St. Gallen, Sankt Gallen
- Ege University Medicine Faculty, Izmir, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided